CLINICAL TRIAL: NCT04169126
Title: Topography Staging and Dual Phase Image Quantification of Tau PET in Cognitive Impairment Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201801834A0
Record Dates: First submitted 2019-11-04; First posted 2019-11-19 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Alzheimer's Disease
Keywords: Dementia; Tau PET scan; Tau neurofibrillary tangles; Amyloid deposition
MeSH Terms: conditions — Alzheimer Disease; Dementia; Amyloidosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F-18-PMPBB3 (Experimental): F-18-PMPBB3 imaging
  Interventions: Drug: F-18 PMPBB3

INTERVENTIONS:
Drug: F-18 PMPBB3 — The study will enroll 200 patients with prodromal AD and AD dementia and 100 normal controls, men and women aged 55-80 years across core clinical criteria of prodromal AD and mild AD dementia based on IWG-2 criteria.

SUMMARY:
A second-generation tau PET image tracer 18F-PM-PBB3 (APN-1607 or MNI-958) has been developed by National Institute of Radiological Sciences. The new tracer solved the off-target binding issue. This study will evaluate new quantitative methods with PMPBB3, by utilized dual phase scanning protocol to extract blood flow and Tau protein binding information, to evaluate appropriate reference brain regions, to improve the normalization efficiency of brain imaging, and to establish a brain template image analysis platform.

DETAILED DESCRIPTION:
Dementia is the top issue in the aging society. Aging population also has its negative implications for the global economy. Effective diagnosis and treatment of dementia is important. Alzheimer's disease accounts for more than 60% of dementia. The main pathological features are the amyloid deposition and Tau neurofibrillary tangles. Currently, our understanding for these misfolded proteins and dementia is limited. There is a need for development of new imaging biomarkers to help clarify the pathophysiology of dementia. In recent years, molecular imaging technology has developed rapidly. In addition to amyloid imaging tracer have been put into clinical use, Tau protein imaging biomarkers have also entered clinical research. However, the tau protein within the patient's brain is not evenly distributed. And the amount of the Tau protein radioactivity is not simply correlate to dementia disease staging. In addition, the problem of off-target binding of the first generation of tracers has yet to be resolved. Recently a second-generation tau PET image tracer 18F-PM-PBB3 (APN-1607 or MNI-958) has been developed by National Institute of Radiological Sciences. The new tracer solved the off-target binding issue. This study will evaluate new quantitative methods with PMPBB3, by utilized dual phase scanning protocol to extract blood flow and Tau protein binding information, to evaluate appropriate reference brain regions, to improve the normalization efficiency of brain imaging, and to establish a brain template image analysis platform. The investigators will evaluate the relationship between Tau protein uptake pattern and disease classifications, and the correlation between Tau protein neurofibrillary tangles and amyloid deposition, and the correlation between MRI and glucose brain connectivity. Finally, to understand the pathophysiology of Tau protein in dementia disease.

ELIGIBILITY:
Inclusion Criteria:

1.1 All subjects

1. Age between 55-80 years
2. Written informed consent must be obtained before any assessment is performed.
3. Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year or, if they are of child-bearing potential, must commit to use a barrier contraception method for the duration of the study.
4. Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method for male subjects for the study duration.
5. Male subjects must not donate sperm for the study duration.
6. Willing to undergo repeated MRIs and at least two PET scans.

1.2 Patient with Prodromal AD or AD dementia

1. Patients fulfill the criteria of prodromal AD or AD dementia based on IWG-2 criteria
2. Able to provide written informed consent with reliable carer in AD population. The participant should have reading ability OR 6/more years of formal education OR with working experiences.

1.3 Cognitive normal control

1. Cognitive unimpaired individual is defined as normal control in this study. Cognitive un-impaired normal control is defined as cognitive performance in the non-impaired range for that individual, defined as not mild cognitive impairment or demented).
2. The normal control should have their clinical dementia rating score 0
3. Cognitive Ability Screening Instrument (CASI) scores rated >50 percentile.

Exclusion Criteria:

1. Already receive outpatient clinic follow-ups with diseases that may affect the cognitive evaluation or presentation that include but not limited to Parkinsonism, Parkinson's disease dementia, schizophrenia, major depression, epilepsy, alcohol or drug abuse, major head trauma with consciousness loss
2. Severe progressive or unstable systemic disease that may interfere with the follow-up and test results. These included but not limited to cancer in the past 5 years, end stage renal or liver dysfunction, clinical significant myocardial infarction (New York Heart Association Functional Classification III-IV), Active disease that received admission in the past one year and unstable angina. Other diseases that were not listed but may interfere with the follow-up or test will be judged by the principle investigator.
3. Any treatment that suggests any of the aforementioned disease will be excluded.
4. Depression with ongoing diagnosis and treatment, suicide idea or suicide behavior in the past 6 months.
5. Contraindications or previously failure for receiving brain magnetic resonance imaging or PET scan.
6. History of risk factors for torsades de pointes (a cardiac dysrhythmia associated with sudden death) or taking medications known to prolong the QT interval.
7. Have an ECG obtained prior to the 18F-PM-PBB3 PET scan that in the opinion of the investigator is clinically significant regarding the subject's participation in the study.
8. Pregnant, lactating or breastfeeding.
9. Patients with severe liver disease (such as ALT > 3x upper limit of normal).

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Tau Distribution Among Normal, Prodromal AD and AD Dementia Subjects Measured by Standardized Uptake Value Ratio (SUVR) as Assessed by 18F-PM-PBB3 tau PET Scan. | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital,Linkou, Taoyuan, Guishan Dist, Taiwan